CLINICAL TRIAL: NCT01400412
Title: A Phase 2b, Double-Blind, Placebo-Controlled, Exploratory Randomized Trial to Determine the Bone, Immunologic, Virologic, and Neurocognitive Effects of a Novel Maraviroc-Containing Antiretroviral Regimen in Treatment-Naïve Patients Infected With R5-Tropic HIV-1
Brief Title: Bone, Immunologic, and Virologic Effects of a Antiretroviral Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5303; 1U01AI068636 (NIH)
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Results first posted 2015-07-15 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Darunavir; Ritonavir; Tenofovir; Emtricitabine; Maraviroc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MVC Arm: DRV/r + MVC + FTC + TDF placebo (Experimental): Darunavir 800 mg PO QD + Ritonavir 100 mg PO QD + Maraviroc 150 mg PO QD + Emtricitabine 200 mg PO QD + Placebo for Tenofovir disoproxil fumarate PO QD
  Interventions: Drug: Darunavir; Drug: Ritonavir; Drug: Emtricitabine; Drug: Placebo for Tenofovir disoproxil fumarate; Drug: Maraviroc
- TDF Arm: DRV/r + TDF + FTC + MVC placebo (Experimental): Darunavir 800 mg PO QD + Ritonavir 100 mg PO QD + Emtricitabine 200 mg PO QD + Tenofovir disoproxil fumarate 300 mg PO QD + Placebo for Maraviroc PO QD
  Interventions: Drug: Darunavir; Drug: Ritonavir; Drug: Tenofovir disoproxil fumarate; Drug: Emtricitabine; Drug: Placebo for Maraviroc

INTERVENTIONS:
Drug: Darunavir — Darunavir was administered orally once a day as two 400 mg tablets with food. When the 800 mg formulation tablet became available, it was substituted for the two 400 mg tablet.
  Other Names: Prezista; TMC-114; DRV
Drug: Ritonavir — Ritonavir was administered orally together with darunavir as one 100 mg tablet once daily with food.
  Other Names: Norvir; RTV
Drug: Tenofovir disoproxil fumarate — Tenofovir disoproxil fumarate was administered orally as one 300 mg tablet once a day.
  Other Names: Viread; TDF
  Arms: TDF Arm: DRV/r + TDF + FTC + MVC placebo
Drug: Emtricitabine — Emtricitabine was administered orally once a day as one 200 mg capsule.
  Other Names: Emtriva; FTC; Coviracil
Drug: Placebo for Tenofovir disoproxil fumarate — Placebo for tenofovir disoproxil fumarate was administered orally once a day as one tablet.
  Arms: MVC Arm: DRV/r + MVC + FTC + TDF placebo
Drug: Placebo for Maraviroc — Placebo for maraviroc was administered orally once a day as one tablet.
  Arms: TDF Arm: DRV/r + TDF + FTC + MVC placebo
Drug: Maraviroc — Maraviroc was administered orally once a day as one 150 mg tablet.
  Other Names: Celesentri; Selzentry
  Arms: MVC Arm: DRV/r + MVC + FTC + TDF placebo

SUMMARY:
The main purpose of this study was to compare the effects on bones of the following two drug combinations:

* maraviroc (MVC), emtricitabine (FTC), plus darunavir/ritonavir (DRV/r)
* tenofovir (TDF) plus emtricitabine (FTC) plus darunavir/ritonavir (DRV/r)

Additional study objectives were the following:

* To see how the drug combinations affect the brain and kidneys.
* To see how well the drug combinations lower the HIV viral load.
* To see how safe the drug combinations are, how well people are able to take the study drug combinations, and how well their immune systems respond to the study drugs.

DETAILED DESCRIPTION:
There are now several HIV treatment options for a person with HIV infection who has not yet been treated. Most people who receive treatment and take their medications as directed have a good result. This is usually determined by measuring the amount of HIV in the blood (viral load). The best response is when HIV cannot be found (less than 50 copies/mL) in the blood. However, it has recently become clear that some people with HIV who are receiving effective HIV drugs continue to have more health problems than people without HIV infection. Sometimes, there is damage to organs in the body, including bone, kidneys, and the brain.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* No evidence of exclusionary resistance mutations defined as evidence of any major NRTI mutation according to the current IAS list of HIV-1 Resistance Mutations Associated with Drug Resistance, or any DRV RAMs (refer to the A5303 PSWP for a list of these mutations) on any genotype; or evidence of significant NRTI or DRV resistance on any phenotype performed at any time prior to study entry. NNRTI-associated resistance mutations were not exclusionary.
* ARV drug-naïve, defined as </=10 days of ART at any time prior to study entry, except in the instances defined in section 4.1.3 of the protocol.
* R5-only tropism based on Trofile testing performed within 90 days prior to study entry.
* Screening HIV-1 RNA >1000 copies/mL obtained within 90 days prior to study entry by any FDA-approved test for quantifying HIV-1 RNA at any laboratory that has a CLIA certification or its equivalent.
* Known hepatitis C virus (HCV) antibody status (performed at any laboratory that had a CLIA certification or its equivalent).
* Certain laboratory values obtained within 60 days prior to study entry, as defined in section 4.1.7 of the protocol.
* For women of reproductive potential, negative serum or urine pregnancy test with a sensitivity of ≤25 mIU/mL within 72 hours prior to study entry.
* Female subjects of reproductive potential, who were participating in sexual activity that could lead to pregnancy, must agree to use at least one reliable method of contraception (as defined in section 4.1.9.1 of the protocol) while receiving the study drugs and for 6 weeks after stopping the medications.
* Female subjects who were not of reproductive potential or whose male partner(s) had azoospermia were eligible to take study drugs without the use of contraceptives.
* Ability and willingness of subject or legal guardian/representative to give written informed consent.
* Willingness to undergo neuropsychological testing.
* DXA scan performed after confirmation of the subject's eligibility by Trofile testing but no more than 4 weeks prior to randomization.

Exclusion Criteria:

* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry.
* New use of hormonal therapies within 6 months prior to study entry. (Stable therapy for ≥6 months was permitted.)
* New use of oral contraceptive pills (OCPs) in the past 3 months. (Stable therapy for ≥3 months was permitted.)
* Any oral, intravenous, or inhaled steroids within 30 days prior to study entry. (Intranasal steroids and topical corticosteroids were allowed.)
* Known allergy/sensitivity to study drugs or their formulations. (A history of sulfa allergy was not an exclusionary condition.)
* Known hypersensitivity to soy lecithin.
* Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or was clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry. (Oral candidiasis, vaginal candidiasis, mucocutaneous herpes simplex, and other minor illnesses (as judged by the site investigator) were not exclusionary conditions.)
* Requirement for any current medications that were prohibited with any study drugs. (Prohibited medications must be discontinued at least 30 days prior to entry. Refer to the A5303 PSWP for a list of prohibited medications.)
* The presence of decompensated cirrhosis.
* A history of or current, active HBV infection defined as positive hepatitis B surface antigen test (or positive HBV DNA in subjects with isolated HBcAb positivity, defined as negative HBsAg, negative HBsAb, and positive HBcAb) at screening.
* Current or prior use of biphosphonates, teriparatide, raloxifene, or denosumab.
* Weight >300 lbs (exceeds weight limit of DXA scanners).
* History after 18 years of age of fracture of the spine, hip, wrist, or other site thought to be related to osteoporosis or bone fragility.
* Currently breastfeeding.
* Any active psychiatric illness including schizophrenia, severe depression, or severe bipolar affective disorder that, in the opinion of the investigator, could confound the analysis of the neurological examination or neuropsychological test results.
* Active drug or alcohol abuse that, in the investigator's opinion, could prevent compliance with study procedures or confound the analysis of study endpoints.
* Active brain infection (except for HIV-1), fungal meningitis, toxoplasmosis, central nervous system (CNS) lymphoma, brain neoplasm, or space-occupying brain lesion requiring acute or chronic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babafemi Taiwo, MBBS, MD, Study Chair — Northwestern University CRS
Locations (38):
- United States (37):
  - 31788 Alabama CRS, Birmingham, Alabama
  - University of Southern California (1201), Los Angeles, California
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Ucsd, Avrc Crs (701), San Diego, California
  - Ucsf Aids Crs (801), San Francisco, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - University of Colorado Denver ATN CRS (33022), Denver, Colorado
  - Georgetown University CRS (GU CRS) (1008), Washington D.C., District of Columbia
  - Children's National Med. Ctr. ATN CRS (33003), Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS (901), Miami, Florida
  - Univ. of South Florida (USF) College of Medicine ATN CRS (33001), Tampa, Florida
  - The Ponce de Leon Center CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - IHV Baltimore Treatment CRS (4651), Baltimore, Maryland
  - 201 Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Washington U CRS (2101), St Louis, Missouri
  - Cooper Univ. Hosp. CRS (31476), Camden, New Jersey
  - Columbia Physicians and Surgeons CRS (30329), New York, New York
  - Trillium Health ACTG CRS (1108), Rochester, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (31787), Rochester, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Moses H. Cone Memorial Hospital CRS (3203), Greensboro, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - Metro Health CRS (2503), Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Hops. of Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - The Miriam Hospital ACTG CRS (2951), Providence, Rhode Island
  - St. Jude Children's Research Hosp. ATN CRS (33016), Memphis, Tennessee
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee
  - Peabody Health Center CRS (31443), Dallas, Texas
  - Houston AIDS Research Team CRS (31473), Houston, Texas
  - Texas Childrens Hospital ATN CRS (33018), Houston, Texas
  - University of Washington AIDS CRS (1401), Seattle, Washington
- Puerto Rico-AIDS CRS (5401), San Juan, Puerto Rico

REFERENCES:
- [Derived] Taiwo BO, Chan ES, Fichtenbaum CJ, Ribaudo H, Tsibris A, Klingman KL, Eron JJ, Berzins B, Robertson K, Landay A, Ofotokun I, Brown T; AIDS Clinical Trials Group A5303 Study Team. Less Bone Loss With Maraviroc- Versus Tenofovir-Containing Antiretroviral Therapy in the AIDS Clinical Trials Group A5303 Study. Clin Infect Dis. 2015 Oct 1;61(7):1179-88. doi: 10.1093/cid/civ455. Epub 2015 Jun 9. PMID 26060295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A5303 opened under version 1.0 on 12/4/11, and the first participant was enrolled on 1/17/12. Accrual to the study closed on 6/12/13, with a total of 262 participants enrolled at 38 sites
Groups:
- MVC Arm (DRV/r + MVC + FTC + TDF Placebo): Darunavir 800 mg PO QD + Ritonavir 100 mg PO QD + Maraviroc 150 mg PO QD + Emtricitabine 200 mg PO QD + Placebo for Tenofovir disoproxil fumarate PO QD
  Darunavir: Darunavir was administered orally once a day as two 400 mg tablets with food. When the 800 mg formulation tablet became available, it was substituted for the two 400 mg tablet.
  Ritonavir: Ritonavir was administered orally together with darunavir as one 100 mg tablet once daily with food.
  Emtricitabine: Emtricitabine was administered orally once a day as one 200 mg capsule.
  Placebo for Tenofovir disoproxil fumarate: Placebo for tenofovir disoproxil fumarate was administered orally once a day as one tablet.
- TDF Arm (DRV/r + TDF + FTC + MVC Placebo): Darunavir 800 mg PO QD + Ritonavir 100 mg PO QD + Emtricitabine 200 mg PO QD + Tenofovir disoproxil fumarate 300 mg PO QD + Placebo for Maraviroc PO QD
  Darunavir: Darunavir was administered orally once a day as two 400 mg tablets with food. When the 800 mg formulation tablet became available, it was substituted for the two 400 mg tablet.
  Ritonavir: Ritonavir was administered orally together with darunavir as one 100 mg tablet once daily with food.
  Tenofovir disoproxil fumarate: Tenofovir disoproxil fumarate was administered orally as one 300 mg tablet once a day.
  Emtricitabine: Emtricitabine was administered orally once a day as one 200 mg capsule.
  Placebo for Maraviroc: Placebo for maraviroc was administered orally once a day as one 150 mg tablet.
Period: Overall Study
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Started | 130 | 132
Completed | 120 | 115
Not Completed | 10 | 17
Not completed — Lost to Follow-up | 4 | 7
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Unable to complete | 3 | 3
Not completed — Never started study treatment | 0 | 3

BASELINE CHARACTERISTICS:
Population: Participants who started study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo) | Total
Number analyzed (Participants) | 130 | 129 | 259
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [26 to 42] | 33 [26 to 42] | 33 [26 to 42]
Age, Customized [Number; unit: participants]
  18-29 Years | 49 | 48 | 97
  30-39 Years | 40 | 41 | 81
  40-49 Years | 26 | 24 | 50
  >=50 Years | 15 | 16 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 115 | 120 | 235
Race/Ethnicity, Customized [Number; unit: participants]
  White non-Hispanic | 57 | 59 | 116
  Black non-Hispanic | 45 | 33 | 78
  Hispanic (regardless of race) | 24 | 34 | 58
  Asian, Pacific Islander | 2 | 1 | 3
  American Indian, Alaskan Native | 0 | 1 | 1
  More than one race | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 127 | 127 | 254
  Puerto Rico | 3 | 2 | 5
CD4 count [Median (Inter-Quartile Range); unit: cells/mm^3] | 389 [295 to 496] | 392 [290 to 518] | 390 [294 to 517]
HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] | 4.59 [3.91 to 5.07] | 4.47 [4.02 to 4.91] | 4.50 [3.97 to 5.00]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density (BMD)
Description: The primary endpoint is the percent change in bone mineral density (BMD) at total hip (as measured by DXA scan) from baseline (week 0) to week 48.
Time Frame: Week 0, week 48
Population: The primary analysis was as-treated which included only participants with total hip BMD measurements available at both week 0 and week 48 who remained on their randomized MVC or TDF component by the time week 48 measurement was taken without an interruption of treatment of more than 10 weeks.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 115 | 109
percentage change | -1.51 [-2.93 to -0.11] | -2.40 [-4.30 to -1.32]
Statistical Analysis 1: Comparison: MVC Arm (DRV/r + MVC + FTC + TDF Placebo) vs TDF Arm (DRV/r + TDF + FTC + MVC Placebo); The null hypothesis is that there is no difference between the two arms in the percent of total hip BMD change from baseline to week 48; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Two-sided p-value without adjustment for multiple testing, interpreted at the 5% nominal level of significance; Stratified Wilcoxon rank sum test stratified by age (<30 and >=30 years)

2. Secondary Outcome: Percent Change in Lumbar Spine Bone Mineral Density (BMD)
Description: The percent change in bone mineral density (BMD) at lumbar spine (as measured by DXA scan) from baseline (week 0) to week 48.
Time Frame: Week 0, week 48
Population: As-treated analysis included only participants with available data at both baseline and week 48 who remained on their randomized MVC or TDF component by the time week 48 DEXA measurement was taken without an interruption of treatment for more than 10 weeks.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 114 | 108
percentage change | -0.88 [-2.93 to 1.30] | -2.35 [-4.25 to -0.45]

3. Secondary Outcome: Change in CD4 Count From Baseline to Week 24
Description: Change in CD4 count from baseline (week 0) to week 24
Time Frame: Week 0, week 24
Population: Change in total CD4 count is analyzed in the same as-treated population as in the primary as-treated analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 115 | 109
cells/mm^3 | 165 [75 to 245] | 127 [35 to 225]

4. Secondary Outcome: Change in CD4 Count From Baseline to Week 48
Description: Change in CD4 count from baseline (week 0) to week 48
Time Frame: Week 0, week 48
Population: Change in total CD4 count is analyzed in the same as-treated population as in the primary as-treated analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 117 | 111
cells/mm^3 | 234 [131 to 327] | 188 [94 to 304]

5. Secondary Outcome: CD8+ T-cell Change From Baseline to Week 48
Description: CD8+ T-cell change from baseline to week 48
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: cell/mm^3
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 117 | 111
cell/mm^3 | -6 [-252 to 175] | -109 [-340 to 59]

6. Secondary Outcome: Percentage Change in Expression of CD38+/HLA-DR+ on CD4+ T Cells From Baseline to Week 48
Description: percentage change is define as [ (week 48 - week 0) / week 0 ] * 100%
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 115 | 108
percentage change | -52.1 [-60.8 to -34.4] | -48.6 [-65.3 to -31.0]

7. Secondary Outcome: Percentage Change in Expression of CD38+/HLA-DR+ on CD8+ T Cells From Baseline to Week 48
Description: percentage change is defined as [ (week 48 - week 0) / week 0 ] * 100%
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | MVC Arm: DRV/r + MVC + FTC + TDF Placebo | TDF Arm: DRV/r + TDF + FTC + MVC Placebo
Number analyzed (Participants) | 115 | 108
percentage change | -59.5 [-70.5 to -43.5] | -60.9 [-71.3 to -49.4]

8. Secondary Outcome: Percent Change in Expression of CD28+/CD57+ on CD8+ T Cells From Baseline to Week 48
Description: percentage change is define as [ (week 48 - week 0) / week 0 ] * 100%
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 115 | 108
percentage change | -9.1 [-24.2 to 9.1] | -11.2 [-29.3 to 16.2]

9. Secondary Outcome: Percent Change in Expression of CD57+ on CD8+ T Cells From Baseline to Week 48
Description: percentage change is define as [ (week 48 - week 0) / week 0 ] * 100%
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 115 | 108
percentage change | -3.5 [-16.9 to 6.5] | -4.6 [-18.4 to 6.6]

10. Secondary Outcome: Percent Change in Expression of CD28+ on CD8+ T Cells From Baseline to Week 48
Description: percentage change is define as [ (week 48 - week 0) / week 0 ] * 100%
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 115 | 108
percentage change | 11.9 [-6.0 to 37.0] | 14.0 [-2.6 to 38.4]

11. Secondary Outcome: Percent Change in Expression of RANKL+ on CD8+ T Cells From Baseline to Week 48
Description: percentage change is defined as [ (week 48 - week 0) / week 0 ] * 100%
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 115 | 108
percentage change | -20.7 [-54.9 to 45.8] | -17.0 [-52.1 to 35.4]

12. Secondary Outcome: Change in Levels of IL-6 From Baseline to Week 48
Description: Change in levels of Interleukin 6 (IL-6) from baseline to week 48
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 116 | 107
pg/ml | -0.21 [-0.91 to 0.25] | -0.12 [-0.83 to 0.42]

13. Secondary Outcome: Change in Level of IP-10 From Baseline to Week 48
Description: Change in level of Interferon gamma-induced protein 10 (IP-10) from baseline to week 48
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 116 | 107
pg/ml | -198 [-366 to -91] | -170 [-310 to -97]

14. Secondary Outcome: Change in Levels of sCD163 From Baseline to Week 48
Description: Change in levels of soluble CD163 from baseline to week 48
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 116 | 107
ng/ml | -250 [-469 to -129] | -258 [-458 to -136]

15. Secondary Outcome: Change in Levels of sCD14 From Baseline
Description: Change in levels of soluble CD14 from baseline
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 116 | 107
ng/ml | -103 [-268 to 63] | -10 [-212 to 159]

16. Secondary Outcome: Change in Levels of D-dimer From Baseline
Description: Change in levels of D-dimer from baseline
Time Frame: At weeks 0 and 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 115 | 106
ng/ml | -82 [-210 to -1] | -61 [-211 to -7]

17. Secondary Outcome: Cumulative Probability of Virologic Failure by Week 48
Description: Confirmed virologic failure is defined as confirmed plasma HIV-1 RNA levels > 1000 copies/mL at or after week 16 and before week 24, or confirmed HIV-1 RNA levels> 200 copies/mL at or after week 24. Participants who discontinued the study with an unconfirmed virologic failure (HIV-1 RNA > 1000 copies at 16 weeks or HIV-1 RNA level > 200 copies/mL at or after week 24) are considered as virologic failures at the study visit week of the unconfirmed value. Time to virologic failure is defined as the time from study entry to the planned visit week of the initial failure.
  Product-limit estimates for the survival function were used to estimate the cumulative probability of virologic failure over time and its corresponding 95% confidence interval for each treatment group.
Time Frame: From study treatment initiation to week 48
Population: All participants who started study treatment
Measure: Number (95% Confidence Interval); unit: cumulative probability per 100 persons
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 130 | 129
cumulative probability per 100 persons | 6 [3 to 12] | 5 [2 to 11]

18. Secondary Outcome: Number of Participants Who Experienced Bone Fractures
Description: Number of participants who experienced bone fractures during the study
Time Frame: From study treatment initiation to week 48
Population: All participants who started study treatment
Measure: Number; unit: participants
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 130 | 129
participants | 2 | 2

19. Secondary Outcome: Number of Participants Who Died During the Study
Description: Number of participants who died during the study
Time Frame: From study treatment initiation to week 48
Population: All participants who started study treatment
Measure: Number; unit: participants
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 130 | 129
participants | 0 | 0

20. Secondary Outcome: Number of Participants Who Developed Grade 3 or 4 Primary Adverse Events
Description: Grade 3 or 4 primary adverse events includes primary signs/symptoms, primary laboratory abnormalities, or primary diagnoses.
  See DAIDS AE Grading Table Version 1.0, Dec 2004 (Clarification, Aug 2009)
Time Frame: From study treatment initiation to week 48
Population: All participants who initiated study treatment
Measure: Number; unit: participants
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Number analyzed (Participants) | 130 | 129
participants | 16 | 22

ADVERSE EVENTS:
Time Frame: week 0 to week 48
Description: Adverse events from participants' first study treatment date to off study date. See DAIDS AE Grading Table Version 1.0, Dec 2004 (Clarification, Aug 2009). All targeted events (see protocol 6.3.4), grade >=3 signs/symptoms or laboratory toxicities, or any adverse events that led to a change in study treatment were required to be recorded.
Arm/Group | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo)
Serious Adverse Events (participants affected / at risk) | 10/130 | 4/129
Other Adverse Events (participants affected / at risk) | 101/130 | 78/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) (N=130) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo) (N=129)
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MVC Arm (DRV/r + MVC + FTC + TDF Placebo) (N=130) | TDF Arm (DRV/r + TDF + FTC + MVC Placebo) (N=129)
Alanine aminotransferase increased (Investigations) | 12 | 15
Aspartate aminotransferase increased (Investigations) | 12 | 10
Blood cholesterol increased (Investigations) | 60 | 39
Blood creatinine increased (Investigations) | 3 | 8
Blood glucose decreased (Investigations) | 7 | 5
Blood glucose increased (Investigations) | 12 | 9
Blood phosphorus decreased (Investigations) | 27 | 24
Blood sodium decreased (Investigations) | 10 | 11
Low density lipoprotein increased (Investigations) | 46 | 26
Neutrophil count decreased (Investigations) | 13 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.